CLINICAL TRIAL: NCT04084587
Title: Visual Rehabilitation Through Acoustic Biofeedback With Retimax Vision Trainer in Patients With Advanced Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Gian Maria Cavallini, Associate Professor, Head of Ophthalmology, Director, School of Specialization in Ophthalmology, University of Modena and Reggio Emilia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 968/2018/DISP/AOUMO
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Macular Degeneration Advanced; Macular Degeneration, Senile; Macular Degeneration, Dry; Macular Scar; Macular Degeneration Nonexudative
Keywords: Rehabilitation; Biofeedback; Retimax Vision Trainer; Age-Related Macular Degeneration; Age-Related Maculopathy; Maculopathies, Age-Related; Retinal Degeneration; Evoked Potentials, Visual
MeSH Terms: conditions — Macular Degeneration, Age-Related, 2; Geographic Atrophy; Macular Degeneration; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Group A: 15 patients rehabilitated with Retimax Vision Trainer, 10 consecutive sessions of 8 minutes each, performed twice a week in the best eye.
  Group B: 9 patients control group without rehabilitation.
  Given the need for constancy and collaboration on the part of the patient, these are allocated to the group of treaties or to the controls based on the fact that they declare themselves more or less available: patients who have transport problems, who live farther away or who in any case they cannot guarantee their presence twice a week, they are allocated to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated Group (Experimental): Group A: 15 patients rehabilitated with Retimax Vision Trainer, 10 consecutive sessions of 8 minutes each, performed twice a week in the best eye.
  Exams performed before and after treatment:
  * BCVA (ETDRS)
  * Reading speed (MNREAD)
  * Contrast sensitivity (Pelli-Robson)
  * Microperimetry and analysis of fixation (OCT-SLO OPTOS)
  * QoL (VFQ-25)
  Interventions: Device: Retimax Vision Trainer
- Control Group (No Intervention): Group B: 9 patients control group without rehabilitation.
  Exams performed twice, at the same time interval elapsed for the treated group:
  * BCVA (ETDRS)
  * Reading speed (MNREAD)
  * Contrast sensitivity (Pelli-Robson)
  * QoL (VFQ-25)

INTERVENTIONS:
Device: Retimax Vision Trainer — The Retimax Vision Trainer is an innovative method that aims to increase visual function in patients with eye diseases of various origins and nature, allowing the patient to exploit and optimize their residual visual potential. It is aimed at patients with visual impairments of different origins and severity, such as campimetric deficits, low vision of central origin, degenerative retinal diseases, amblyopia. (1,2) It consists of a device for recording bioelectrical responses evoked during the perception of structured visual stimuli and the control of the same by the patient through a sound biofeedback mechanism. This results in an increase in visual capacity, exploiting neuronal plasticity through the activation of alternative neuronal circuits.
  Arms: Treated Group

SUMMARY:
At present there are no real therapies able to improve visual performance in patients with age-related macular degeneration, atrophic type. The aim of the study is to verify whether with rehabilitation sessions with Retimax Vision Trainer it is possible to teach the maculopathic patient to exploit the extrafoveal areas of the retina, not affected by atrophy, resorting to an eccentric vision that compensates for the foveal one, thus obtaining a improvement of visual outcomes (far and near vision capacity, sensitivity to contrast to reading, reading speed, fixation capacity and overall quality of life of the visually impaired patient suffering from atrophic senile maculopathy (AMD)). To do this, the study design was conceived as a non-randomized prospective comparative and involves the formation of two groups of patients: a group A of 15 patients who will be rehabilitated with Retimax and a group B of 15 patients who will not be rehabilitated, but only re-evaluated at the same distance of time that will elapse for group A. Eligible patients are affected by atrophic AMD with unstable fixation and better vision in the eye between 1/10 and 4/10 in the absence of other serious eye diseases. As there is currently no real therapy capable of improving visual performance, the demonstration of the positive effect of the visual rehabilitation program with Retimax in patients suffering from atrophic macular degeneration may encourage a wider use of this method. The patient could benefit from a non-invasive, repeatable and cost-effective procedure.

DETAILED DESCRIPTION:
Study typology:

prospective, non-randomized, monocentric, comparative study. There is no agreement between promoter and clinical center. There is no agreement between promoter and financier: the study has no funding.

Background:

The Retimax Vision Trainer is an innovative method that aims to increase visual function in patients with eye diseases of various origins and nature, allowing the patient to exploit and optimize their residual visual potential. It is aimed at patients with visual impairments of different origins and severity, such as campimetric deficits, low vision of central origin, degenerative retinal diseases, amblyopia.

It consists of a device for recording bioelectrical responses evoked during the perception of structured visual stimuli and the control of the same by the patient through a sound biofeedback mechanism. This results in an increase in visual capacity, exploiting neuronal plasticity through the activation of alternative neuronal circuits. The device has already been used in clinical practice at the AOU Modena for about a year precisely with the indication of rehabilitation in the visually impaired patients: therefore the current indication includes that of the study in question. Subjects with central low vision, such as those with advanced AMD, tend to develop independently an eccentric fixation area (PRL or Preferred Retinal Locus) which is generally found on the horizontal meridian of the fovea, mainly on the interpapillo-macular beam.

However, this situation represents an obstacle because it does not allow a continuous vision, for example preventing reading and writing which would require a strip of healthy retinal tissue long enough to allow the simultaneous viewing of at least 10-12 words.

For this reason patients suffering from central hypovision can benefit from rehabilitative programs with bio-feedback mechanism that teach to move the eye to translate the PRL from the central degenerated area to an adjacent healthy area large enough to allow reading / writing . This leads to the formation of a TRL, Trained Retinal Locus, which is generally found in the upper parafoveal area (projected in the lower part of the visual field to be more functional for daily activities such as, for example, reading).

The most widespread rehabilitation method is stimulation with bio feedback. Each rehabilitation cycle is customized but generally involves twice-a-week sessions in the first five weeks for the creation of the TRL followed by maintenance sessions on a fortnightly basis. At the end of the rehabilitation period it is always advisable to send the patient to the test of the most appropriate aids. Rehabilitation sessions are performed only on the eye with better visual acuity since binocular fixation is determined by the eye with better vision than by the dominant eye.

Purpose:

The purpose of the study is to evaluate the effectiveness of rehabilitation through acoustic biofeedback with Retimax Vision Trainer in patients with low vision suffering from age-related macular degeneration in the advanced phase, in order to demonstrate the positive effect that this treatment has on far and near vision, on the contrast sensitivity, on the reading speed, on the ability to fix and on the overall quality of life of the patient. We will therefore try to highlight the quantitative variation of these parameters between pre and post rehabilitation by comparing two groups of patients, one subjected to rehabilitation and one not and we will try to understand if this variation is significant.

Group A: 15 patients rehabilitated with Retimax Vision Trainer, 10 consecutive sessions of 8 minutes each, performed twice a week in the best eye.

Group B: 15 patients control group without rehabilitation.

Given the need for constancy and collaboration on the part of the patient, these are allocated to the group of treated or to the controls based on the fact that they declare themselves more or less available: patients who have transport problems, who live farther away or who in any case they cannot guarantee their presence twice a week, they are allocated to the control group.

Materials and methods:

Patients will be enrolled during visits to the maculopathy outpatient clinic that follows patients at the end of the cycle for intravitreal injections with anti-VEGF. The enrolled maculopathies are atrophic, therefore in the study there will be both patients with advanced forms of maculopathy who have exhausted the role of anti-VEGF, but also patients with pure atrophic forms who have never performed intravitreal. Therefore, enrollment is independent of the administration of anti-VEGF.

It will be proposed to participate in the study, providing the information sheet and holding an interview explaining the importance of consistency in rehabilitation sessions and what the method consists of. Subsequently consent will be collected. At the signing of the consent, personal data will be collected. The patient will be told that he will be contacted by telephone in the following days to fix the date of the first pre-treatment visit.

Exams performed before and after treatment:

* BCVA (ETDRS)
* Reading speed (MNREAD)
* Contrast sensitivity (Pelli-Robson)
* Microperimetry and analysis of fixation (OCT-SLO OPTOS)
* QoL (VFQ-25)

After the visit, the patient will be contacted by the orthoptists to fix the 10 rehabilitation sessions with Retimax, twice a week. At the end a final post-treatment visit will be repeated, repeating all the exams. At this point we will proceed with statistical analysis, with the help of a biostatisticist, to evaluate the effectiveness of visual rehabilitation.

Statistic analysis The study data are extrapolated from each patient and divided into pre and post-treatment.

The pre-treatment value and the post-treatment value of each single parameter for each individual patient will be compared with each other trying to demonstrate the improvement and the significance of the variation.

For statistical calculations we will use the software R: A language and environment for statistical computing, version 3.3.3, R Foundation for Statistical Computing, Vienna, Austria (http://www.R-project.org/) with the collaboration of a biostatistics expert.

Given the non-normal distribution verified with the Shapiro-Wilk test and the low number, the pre and post treatment values will be compared with the One-sided Wilcoxon Signed Rank Test

Expected results:

* Improvement of fixation capacity and microperimetry
* Improvement of visual acuity, reading speed and contrast sensitivity
* Improvement of sight quality

ELIGIBILITY:
Inclusion Criteria:

Patients were included in the study based on the following criteria:

* Diagnosis of advanced age-related macular degeneration through examination of the fundus oculi and OCT;
* Best corrected visual acuity (BCVA) for far in the best eye between 1/10 and 4/10;
* Collaborating patients with a positive attitude towards a rehabilitation treatment with a bi-weekly commitment.

Exclusion Criteria:

The exclusion criteria from the study are:

* Presence of concomitant retinal or optic nerve pathologies;
* Eye surgery more recent than six months, except for the cataract for which the cut off is fixed at two months;
* Poor collaboration by the patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Far Visual Acuity pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Far Visual Acuity was measured for each eye, with the best refractive correction of visus (BCVA) using Logaritmic Visual Acuity Chart ETDRS, R chart, Precision Vision La Salle Illinois, Usa at 8 feet (2.44m) of distance. The number of letters read by the patient was used for statistical analyzes.
Change in Contrast Sensitivity pre and post treatment | one week before the treatment starts and one week after the treatment stops
  The Contrast Sensitivity was measured for each eye, with the best refractive correction of visus (BCVA) using Pelli-Robson Contrast Sensivity Chart, Precision Vision La Salle Illinois, Usa at 1 m distance. LogSC values were used for statistical analyzes.
Change in Near Visual Acuity pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Near visual acuity was measured for each eye, with the best refractive correction of vision (BCVA) using 35 ± 5 cm MNREAD Acuity Charts, Precision Vision La Salle Illinois, USA, distributed in the Italian version by Carl Zeiss Jena GmbH, Germany.
  This test consists of graphs containing 19 sentences. Each sentence is printed in three lines. The sentences are in different print formats ranging from 1.3 to -0.5 logMAR and each of them is 0.1 logMAR units smaller than the previous sentence (about 80% of the size). Patients read the graphic aloud starting from the largest characters to reach the smallest characters and, simultaneously, the time required for reading and the frequency of errors are recorded.
  Near visual acuity is measured in relation to the smallest character that the patient can read without making significant errors. LogMAR values were used for statistical analyzes.
Change in Reading Speed pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Reading Speed was measured for each eye, with the best refractive correction of vision (BCVA) using 35 ± 5 cm MNREAD Acuity Charts, Precision Vision La Salle Illinois, USA, distributed in the Italian version by Carl Zeiss Jena GmbH, Germany. Each sentence consists of 60 characters, corresponding to 10 words of standard length, considered 6 characters (including the space between one word and another), so that each sentence can be divided into 10 smaller units. Patients read the graphic aloud and, simultaneously, the time required for reading and the frequency of errors are recorded. The maximum reading speed (MRS) was calculated with reference to the time taken by the patient to read the sentence corresponding to his visual acuity for near. Since the number of words in the sentence is fixed, it is possible with a simple proportion to calculate the reading speed expressed in words per minute (WpM). WpM values were used for statistical analyzes.
Change in Score in the Questionnaire "Quality of Life" pre and post treatment | one week before the treatment starts and one week after the treatment stops
  To assess the impact that low vision maculopathy has on daily life, patients were subjected to a National Eye Institute Visual Functioning Questionnaire -25 (NEI VFQ-25) translated into Italian. It is a test composed of 25 questions divided into 3 areas: general health and vision, difficulties in daily activities, response to visual problems. The test was released to the patient who completed it independently; in cases of marked low vision, it can be administered directly by reading aloud. For each response, a score was assigned based on the National Eye Institute's indication for a total variable from 0 to 100. Major final score indicates a better quality of life for the patient. For the statistical analyzes the values of the final score of the test were used.
Change in Retinal sensitivity to microperimetry pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Patients undergo microperimetry to study retinal sensitivity and fixation. The instrument used to perform the microperimetry is the Spectral OCT-SLO combination imaging system, Optos, Dunfermline, Scotland, UK. The Spectral OCT / SLO is an optical acquisition system designed to capture images of the retinal layers (OCT) simultaneously with confocal images of the ocular fondus (SLO). It is mainly used in OCT mode, but has a specific microperimetry program. The instrument is also equipped with built-in lenses used to correct the patient's refraction (from -20.00 to +18.00 D). In our study the sights used are of the Goldmann III type, white in color, with a duration of 200 ms; 28 points were stimulated arranged according to a grid created around the macula with strategy 4.2. An attenuation scale of 20 dB was used with a maximum stimulus intensity of 400asb equal to 0 dB. The fixation target, established at 100 asb, is represented by a circle of the magnitude of a degree.
Change in Fixation in the 2 central degrees pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Patients undergo microperimetry to study retinal sensitivity and fixation. The instrument used to perform the microperimetry is the Spectral OCT-SLO combination imaging system, Optos, Dunfermline, Scotland, UK. The Spectral OCT / SLO is an optical acquisition system designed to capture images of the retinal layers (OCT) simultaneously with confocal images of the ocular fondus (SLO). It is mainly used in OCT mode, but has a specific microperimetry program. The instrument is also equipped with built-in lenses used to correct the patient's refraction (from -20.00 to +18.00 D). In our study the sights used are of the Goldmann III type, white in color, with a duration of 200 ms; 28 points were stimulated arranged according to a grid created around the macula with strategy 4.2. An attenuation scale of 20 dB was used with a maximum stimulus intensity of 400asb equal to 0 dB. The fixation target, established at 100 asb, is represented by a circle of the magnitude of a degree.
Change in Fixation in the 4 central degrees pre and post treatment | one week before the treatment starts and one week after the treatment stops
  Patients undergo microperimetry to study retinal sensitivity and fixation. The instrument used to perform the microperimetry is the Spectral OCT-SLO combination imaging system, Optos, Dunfermline, Scotland, UK. The Spectral OCT / SLO is an optical acquisition system designed to capture images of the retinal layers (OCT) simultaneously with confocal images of the ocular fondus (SLO). It is mainly used in OCT mode, but has a specific microperimetry program. The instrument is also equipped with built-in lenses used to correct the patient's refraction (from -20.00 to +18.00 D).In our study the sights used are of the Goldmann III type, white in color, with a duration of 200 ms; 28 points were stimulated arranged according to a grid created around the macula with strategy 4.2. An attenuation scale of 20 dB was used with a maximum stimulus intensity of 400asb equal to 0 dB. The fixation target, established at 100 asb, is represented by a circle of the magnitude of a degree.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Maria Cavallini, Associate Professor, Principal Investigator — Dipartimento Chirurgico, Medico, Odontoiatrico e di Scienze Morfologiche con interesse Trapiantologico, Oncologico e di Medicina Rigenerativa -UNIMORE- University of Modena and Reggio Emilia
Locations (1):
- Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided